CLINICAL TRIAL: NCT06023381
Title: Sliding Sign in Third-trimester Ultrasound Evaluation of Intra-abdominal Adhesions in Women Undergoing Repeat Cesarean Section
Brief Title: Sliding Sign in Late Trimester Ultrasound Evaluation of Intra-abdominal Adhesions in Women Undergoing Repeat CS
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Al Shirbiny Hamed Esmail, Principal Investigator, Ain Shams Maternity Hospital
Other Study IDs: Sliding Sign
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sliding sign — All women had Transabdominal Ultra-sonography using SAMSUNG WS80 "elite" ultrasound machine during the preoperative examination, using the real-time Transabdominal pelvic features (the relative motion between the maternal abdominal and uterine wall).
  The patient was asked to breathe deeply, accentuating her respiratory movements and the sonographer recorded a video clip in a mid-sagittal plane lateral to umbilicus focus on the infra-umbilical space, to determine whether the structure glided freely in relation to adjacent structures. To be considered as sliding, the structures had to glide easily, one against the other (positive sliding sign); no motion of the structure in question signaled a negative sliding sign.

SUMMARY:
Predicting the presence of severe adhesions may also assist clinically in several ways: first, it allows allocation of more complicated surgeries to experienced surgeons; second, the surgeons can plan and prepare better for the surgery if they know in advance whether they are going to operate a complicated surgery; third, a difficult surgery may be scheduled to be performed in an experienced center, preparing cross match blood units, and alerting the general surgeon and urologist of the potential risk for surgical complications, saving time if intervention is required.

This information can permit preoperative planning by a multidisciplinary team of surgeons and allow the patient to be informed of the potentially high risk of complications.

DETAILED DESCRIPTION:
The incidence of repeat cesarean delivery is on the rise worldwide, approximately 90% of women with a prior cesarean delivery undergo a planned repeat cesarean delivery in their next pregnancy.

Post-cesarean adhesions are a major complication in subsequent surgeries, causing an increased risk for bladder and bowel injury (0.1-0.3%), hemorrhage (0.1-1.4%), infection (0.4-1.6%), and even hysterectomy (0.1-1.4%).

In addition to the risk associated with the pelviabdominal surgical procedure itself, adhesiolysis may result in injury to adjacent viscera, blood loss, and in case of emergency cesarean delivery, to the perinatal adverse outcome associated with delayed delivery of the neonate. This represents a considerable healthcare issue, as it has a significant impact both on the patient, increasing morbidity and mortality, and on healthcare costs. It is therefore important for surgeons to detect patients at high risk of having adhesions.

Women suspected to have severe intra-abdominal adhesions may benefit from appropriate preparation of blood products, better assignment of surgeons, request for preoperative surgical assistance of other medical specialties, and possibly performance of a midline skin incision to enter the peritoneal cavity. It is therefore important for surgeons to detect patients at high risk of having adhesions.

Various means have been proposed to predict adhesions prior to surgery, including analysis of patient characteristics and appearance of the scar, as well as the intraoperative peritoneal adhesion index.

ELIGIBILITY:
Inclusion Criteria:

1. History of previous cesarean section.
2. Gestational age: Full-Term.
3. Scheduled to undergo elective cesarean section.

Exclusion Criteria:

1. Body mass index more than 40 on admission.
2. Abnormal placental invasion.
3. Having known collagen disease.
4. Unplanned or emergency repeated cesarean delivery.
5. History of abdominal surgery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All third trimester pregnant women with a history of previous cesarean section who were admitted for elective caesarian section had Transabdominal Ultra-sound during the preoperative examination, using the real-time Transabdominal ultrasound pelvic features
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
The association between a negative sliding sign and severe adhesions | 24 hours
  through transabdominal ultrasound

SECONDARY OUTCOMES:
The association between a negative sliding sign and operative time | 24 hours
  time from skin incision to delivery of the baby
hemoglobin drop greater than 3 g/dL | 24 hours
  calculated between preoperative and postoperative hemoglobin levels
Urinary Bladder injury | 24 hours
  intraoperative diagnosis or postoperatively
Intestinal injury | 24 hours
  intraoperative diagnosis or postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Rania Gamal, MD, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Faculty of Medicine, Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No